CLINICAL TRIAL: NCT02523157
Title: Wellbeing in Pregnancy: Evaluating an Intervention to Improve Women's Emotional Wellbeing in Pregnancy
Acronym: WiP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: Boots Family Trust (Unknown); Tommy's (Other); Netmums (Unknown); Institute of Health Visiting (Unknown); Royal College of Midwives (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: CityULondon
Record Dates: First submitted 2015-07-29; First posted 2015-08-14 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2015-08

CONDITIONS: Peripartum Period; Mental Health; Pregnant Women
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Wellbeing Plan
  Interventions: Other: Wellbeing Plan
- Control (Active Comparator): Control task. Information about physical health in pregnancy, matched for readability (Flesch score) and length/duration with the Wellbeing Plan
  Interventions: Other: Control task

INTERVENTIONS:
Other: Wellbeing Plan — The Wellbeing Plan is a short self-help leaflet designed to improve emotional wellbeing of women during and after pregnancy by providing information, raising awareness, helping a woman identify her own symptoms, provide coping strategies, and identify key people who can support the woman during this time.
  Arms: Intervention
Other: Control task — Information about physical health in pregnancy, matched for readability (Flesch score) and length/duration with the Wellbeing Plan
  Arms: Control

SUMMARY:
The Wellbeing in Pregnancy (WiP) project is an online pilot randomized controlled trial which aims to evaluate an intervention to improve women's emotional wellbeing in pregnancy.

DETAILED DESCRIPTION:
It is estimated that mental health problems affect 10-20% of postnatal women. Many of these women do not seek help for their mental health for numerous reasons, including lack of awareness about symptoms, available treatments, and stigma. The Wellbeing Plan is a brief self-help leaflet developed by experts in perinatal mental health, and is designed to improve emotional wellbeing of women during and after pregnancy by providing information, raising awareness, helping a woman identify her own symptoms, provide coping strategies, and identify key people who can support the woman during this time. The Wellbeing in Pregnancy project is a online pilot randomized controlled trial which aims to evaluate the efficacy of the Wellbeing Plan in improving women's emotional wellbeing in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 26-38 weeks pregnant
* Sufficient proficiency in English to understand and complete the Wellbeing Plan

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in knowledge and beliefs about perinatal mental health from baseline at 1 month | Baseline to 1 month
  Knowledge and beliefs about perinatal mental health will be measured using a 12-item self-report questionnaire scored on a 5-point Likert scale from 1 = Strongly agree to 5 = Strongly disagree. It has been developed in consultation with the research team and with a parental advisory group. It will explore women's knowledge and beliefs about perinatal mental health problems, including perceived stigma, incidence of psychological distress in the perinatal period, as well as knowledge and beliefs regarding sources of potential support for women.

SECONDARY OUTCOMES:
Changes in mood from baseline at 1 month | Baseline to 1 month
  Small changes in mood will be examined using the UWIST Mood Adjective Checklist (UMACL; Mathews, Jones & Chamberlain, 1990). The UMACL includes 24 mood adjectives. Participants indicate whether each adjective relates to their current mood on a 4-point scale with higher scores indicating stronger mood. It has 3 subscales of tense arousal (8 items), energetic arousal (8 items) and hedonic tone (8 items), which have been confirmed by factor analysis. For this study, the items relating to energetic arousal will be omitted, as energy levels will be affected by the late pregnancy stage/early postpartum period.
Changes in mood from baseline at 6 weeks postpartum | Baseline to 6 weeks postpartum
  Small changes in mood will be examined using the UWIST Mood Adjective Checklist (UMACL; Mathews, Jones & Chamberlain, 1990). The UMACL includes 24 mood adjectives. Participants indicate whether each adjective relates to their current mood on a 4-point scale with higher scores indicating stronger mood. It has 3 subscales of tense arousal (8 items), energetic arousal (8 items) and hedonic tone (8 items), which have been confirmed by factor analysis. For this study, the items relating to energetic arousal will be omitted, as energy levels will be affected by the late pregnancy stage/early postpartum period.
Changes in general psychological health from baseline at 1 month | Baseline to 1 month
  General psychological health will be measured using the CORE-10 (Barkham et al, 2013; Connell & Barkham, 2007).
Changes in general psychological health from baseline at 6 weeks postpartum | Baseline to 6 weeks postpartum
  General psychological health will be measured using the CORE-10 (Barkham et al, 2013; Connell & Barkham, 2007).
Changes in depressive symptoms from baseline at 1 month | Baseline to 1 month
  The Whooley questions (NICE, 2014) will be used to measure clinically relevant depression.
Changes in depressive symptoms from baseline at 6 weeks postpartum | Baseline to 6 weeks postpartum
  The Whooley questions (NICE, 2014) will be used to measure clinically relevant depression.
Changes in general anxiety symptoms from baseline at 1 month | Baseline to 1 month
  The GAD-2 (Kroenke et al, 2007) will be used to measure clinically relevant anxiety.
Changes in general anxiety symptoms from baseline at 6 weeks postpartum | Baseline to 6 weeks postpartum
  The GAD-2 (Kroenke et al, 2007) will be used to measure clinically relevant anxiety.
Changes in perceived support from baseline at 1 month | Baseline to 1 month
  Perceived support will be measured using the Maternity Social Support Scale (MSSS) (Webster et al, 2000). The MSSS is a 6-item self-report questionnaire rated on a 5-point Likert scale which measures perceived social support in the prenatal period. It examines the woman's relationship with her partner, exploring the nature of the relationship, in addition to perceived support from family and friends.
Changes in perceived support from baseline at 6 weeks postpartum | Baseline to 6 weeks postpartum
  Perceived support will be measured using the Maternity Social Support Scale (MSSS) (Webster et al, 2000). The MSSS is a 6-item self-report questionnaire rated on a 5-point Likert scale which measures perceived social support in the prenatal period. It examines the woman's relationship with her partner, exploring the nature of the relationship, in addition to perceived support from family and friends.
Changes in help-seeking behaviors from baseline at 1 month | Baseline to 1 month
  Help-seeking behaviours will be assessed by asking women if they have spoken to anyone about their feelings, if they have been worried about their mental wellbeing.
Changes in help-seeking behaviors from baseline at 6 weeks postpartum | Baseline to 6 weeks postpartum
  Help-seeking behaviours will be assessed by asking women if they have spoken to anyone about their feelings, if they have been worried about their mental wellbeing.
Changes in knowledge and beliefs about perinatal mental health from baseline to 6 weeks postpartum | Baseline to 6 weeks postpartum
  Knowledge and beliefs about perinatal mental health will be measured using a 12-item self-report questionnaire scored on a 5-point Likert scale from 1 = Strongly agree to 5 = Strongly disagree. It has been developed in consultation with the research team and with a parental advisory group. It will explore women's knowledge and beliefs about perinatal mental health problems, including perceived stigma, incidence of psychological distress in the perinatal period, as well as knowledge and beliefs regarding sources of potential support for women.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Ayers, PhD, Principal Investigator — City, University of London
Locations (1):
- City University London, London, London, United Kingdom

REFERENCES:
- [Background] Barkham M, Bewick B, Mullin T, Gilbody S, Connell J, Cahill J, ... & Evans C. The CORE-10: A short measure of psychological distress for routine use in the psychological therapies. Counselling and Psychotherapy Research, 13(1): 3-13, 2013. doi: 10.1080/14733145.2012.729069
- [Background] Boots Family Trust Alliance. Perinatal Mental Health Experiences of Women and Health Professionals, 2013. Retrieved from: http://www.tommys.org/file/Perinatal_Mental_Health_2013.pdf
- [Background] Boyatzis RE. Transforming qualitative information: thematic analysis and code development. London: Sage; 1998.
- [Background] Connell J, & Barkham M. CORE-10 User Manual, Version 1.1. CORE System Trust & CORE Information Management Systems Ltd, 1-40, 2007.
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Leadsom A, Field F, Burstow P & Lucas C. The 1001 Critical Days: The Importance of the Conception to Age Two Period, 2014. Retrieved from: http://www.andrealeadsom.com/downloads/1001cdmanifesto.pdf
- [Background] Maternal Mental Health Alliance. The Costs of Perinatal Mental Health Problems. London: Centre for Mental Health, 2014.
- [Background] Matthews G, Jones DM, & Chamberlain AG. Refining the measurement of mood: The UWIST Mood Adjective Checklist. British Journal of Psychology 81: 17-42, 1990.
- [Background] NICE. Guideline CG192: Antenatal and Postnatal Mental Health: clinical management and service guidance, 2014. Retrieved from: http://www.nice.org.uk/guidance/cg192/chapter/1-recommendations#recognising-mental-health-problems-in-pregnancy-and-the-postnatal-period-and-referral-2
- [Background] NSPCC. Prevention in Mind. All Babies Count: Spotlight on Perinatal Mental Health, 2013. Retrieved from: http://www.nspcc.org.uk/globalassets/documents/research-reports/all-babies-count-spotlight-perinatal-mental-health.pdf
- [Background] Office for National Statistics. Statistical Bulletin: Births and deaths in England and Wales 2011. Newport: Office for National Statistics, 2012.
- [Background] O'Hara MW, & Swain AM. Rates and risk of postpartum depression - a meta-analysis. International review of psychiatry 8(1): 37-54, 1996.
- [Background] Robertson E, Grace S, Wallington T, Stewart DE. Antenatal risk factors for postpartum depression: a synthesis of recent literature. Gen Hosp Psychiatry. 2004 Jul-Aug;26(4):289-95. doi: 10.1016/j.genhosppsych.2004.02.006. PMID 15234824
- [Background] Webster J, Linnane JW, Dibley LM, Hinson JK, Starrenburg SE, Roberts JA. Measuring social support in pregnancy: can it be simple and meaningful? Birth. 2000 Jun;27(2):97-101. doi: 10.1046/j.1523-536x.2000.00097.x. PMID 11251486
- See also: Guideline CG192: Antenatal and Postnatal Mental Health: clinical management and service guidance. — http://www.nice.org.uk/guidance/cg192/chapter/1-recommendations#recognising-mental-health-problems-in-pregnancy-and-the-postnatal-period-and-referral-2
- See also: Prevention in Mind. All Babies Count: Spotlight on Perinatal Mental Health. — http://www.nspcc.org.uk/globalassets/documents/research-reports/all-babies-count-spotlight-perinatal-mental-health.pdf
- See also: Wellbeing Plan — http://www.bftalliance.co.uk/wellbeing-plan/